CLINICAL TRIAL: NCT03934879
Title: Physical Exercise and Contributors to Academic Performance Among Adolescents With ASD (Fit Club Study)
Acronym: FitClub
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-0185
Record Dates: First submitted 2016-08-08; First posted 2019-05-02 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2020-04

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: One school will receive FitClub intervention. Second school will receive regular school activities.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gateway Academy (Experimental): For this study, Gateway Academy students will participate in the FitClub intervention. They will rotate through each fitness module, which includes spin class, Pilates, strengthening exercises (weight training), basketball, running and rhythm, and cardio fitness. Students will meet five days per week during their first class of the day for 35 minutes and participate in two randomly assigned modules for two week periods. After 2 weeks, they participate in 2 different modules. Resting and peak heart rate (during exercise), calories burned and steps taken will be collected during each session.
  Interventions: Behavioral: FitClub
- Control School (Active Comparator): Other comparable school will be added as a control school, in which regular school activities will be provided.
  Interventions: Other: Regular School Activities

INTERVENTIONS:
Behavioral: FitClub — Participants will rotate through each fitness module, which includes spin class, Pilates, strengthening exercises (weight training), basketball, running and rhythm, and cardio fitness. Students will meet five days per week during their first class of the day for 35 minutes and participate in two randomly assigned modules for two week periods. After 2 weeks, they participate in 2 different modules. Resting and peak heart rate (during exercise), calories burned and steps taken will be collected during each session.
  Arms: Gateway Academy
Other: Regular School Activities — Students will participate in regular school activities.
  Arms: Control School

SUMMARY:
This study, Physical Exercise and Contributors to Academic Performance among Adolescents with Autism Spectrum Disorders (ASD), aims to expand our understanding of the impact of regular physical exercise on improvement in academic performance. The investigators will focus on the use of affordable, portable, and achievable interventions that can be easily shared and incorporated into other academic and home settings. The study will examine the use a regular vigorous exercise program for helping students with ASD reduce body mass index and improve executive function, motor performance, sensory responsiveness, and mood. The investigators propose a collaborative arrangement with an area school to conduct an 18-month exploratory pilot study of 30 middle- and high-school aged students (12 to 18 years old) with ASD, who are returning participants or are new to participating in the Fit Club at Gateway Academy. The investigators expect that the changes elicited by participation in this type of exercise program will support the formation of adult life skills, impacting on long-term quality of life for individuals with ASD and children with other conditions.

DETAILED DESCRIPTION:
Detailed Description: Background:

Individuals with autism spectrum disorders (ASD) typically have social impairment, have difficulty making decisions and problem solving (executive function) and have impaired motor performance. As a result, they are less likely to even live independently, be employed, go to college or get married. Few effective interventions have been found to help with the complex problems of people with ASD who are unable to establish independent lives. The investigators plan to begin the examination of using a regular physically challenging exercise program to support development of executive function (EF) and motor skills among children and young adults with ASD to improve academic behaviors and participation in adult activities.

In addition to having social, EF and motor problems, children and young adults with ASD often participate in limited physical activities, enjoy them less than do typically developing (TD) children, are less motivated to participate in physical activities than TD children, experience weight gain from medications, and encounter problems with reduced physical fitness and obesity. Lack of interest or motivation to exercise may make it difficult for them to comply with daily physical activity recommendations. As a result, these students are less likely to be involved in physical activity, enjoy fewer types of leisure activities, and experience limited relationships with peers, which eventually contribute to lower levels of participation in adult activities.

Benefits of Physical Activity:

Physical exercise has been shown to improve cognitive processes in TD individuals. It has a positive influence on symptoms seen in children and adolescents with ASD, including experiencing reductions in stereotypical behaviors, improved sensory skills and social responsiveness, improved concentration and memory, weight reduction, improved motor skills, improvement in executive function and a reduction in repetitive behaviors. Many of these skills are necessary for adult tasks such as driving, test-taking, employment, and engaging in other purposeful adult activities. The mechanism of improvement in these cognitive functions as a result of physical exercise is thought to be caused by increased cerebral blood flow, up-regulation of neuroprotective growth factors, and the cardiovascular benefits of exercise, which lead to an improvement in the delivery of oxygen and nutrients. It is not clear, however, if the amount of effort during exercise is related to the improvement in cognitive functions.

Participation: Participation in activities is how children and young adults develop an understanding of the expectations of society and gain the physical and social skills needed to function and flourish, it plays an important role in a child's or young adult's social development, and it influences long-term mental and physical health.

Mood: Having ASD may lead to psychosocial impairments, including depression, anxiety, stress, and low self-esteem. For example, Shtayermman (2008) reported that 50% of study participants with Asperger syndrome had made a suicide attempt, while Paquette-Smith, Weiss, and Lunsky (2014) determined that "36% suicide attempt rate reported in their sample of 50 adults with Asperger Syndrome was much higher than the national average of 4.6% over a lifetime in the general population". Using the Depression, Anxiety, and Stress Scale (DASS-21), components of psychosocial well-being will be assessed in this cohort of children during this study.

Sensory Responsiveness: Children and young adults with ASD demonstrate unusual sensory responses to stimuli more frequently than do typically developing peers or those with other developmental disorders. In a study comparing children with and without ASD, atypical sensory responsiveness patterns greater than one standard deviation from the mean were found in up to 95% in children with ASD, compared to 12 to 25% of children without ASD in the various sensory domains.

Gateway Academy: For this study, the investigators will partner with Gateway Academy, a private school that utilizes innovative approaches to learning, physical fitness, and social awareness, and enrolls approximately 55 students of middle to high school age with social and academic challenges, the majority of whom have an ASD diagnosis. Gateway Academy developed a Fit Club fitness program seven years ago modeled after an exercise program developed by Ratey. In addition, a second school, closely matched to Gateway Academy functional levels, has communicated an interest in participating in the second stage of this study.

Methodology:

Each year, 10 to 15 new students join Gateway Academy who have not participated in an organized, mandatory exercise intervention (Fit Club). With this study, the investigators plan to examine the impact of the Fit Club intervention by comparing students new to the Fit Club intervention throughout the school year, and also by tracking returning students on a range of factors, including BMI, executive function, motor skills, sleep patterns, and classroom behaviors.

The investigators propose to conduct an 18-month exploratory pilot study of 30 middle- and high-school aged students (12 to 18 years old) with ASD, who participate in, or are new to participating in the Fit Club at Gateway Academy. Engagement in exercise and response to exercise will be constantly monitored for participants. Other participant data will be collected three times, once at baseline, at the end of the school year, and at the beginning of the next school year.

The investigators will adhere to the Fit Club fitness program protocol. All students will rotate through each fitness module, which includes spin class, Pilates, strengthening exercises (weight training), basketball, running and rhythm, and cardio fitness. Students will meet five days per week during their first class of the day for 35 minutes and participate in two randomly assigned modules for two week periods. After 2 weeks, they participate in 2 different modules.

Study Objectives:

Objective 1: To determine how students new to the fitness program compare to their returning peers in BMI, executive function, sensory responsiveness, motor skills, mood, and activity participation.

Objective 2: To quantify the changes in BMI, executive function, sensory responsiveness motor skills, and mood after participation in a fitness program after one and two semesters for new and returning students.

Objective 3: To determine if greater physical effort is correlated with greater improvement in BMI, executive function, sensory responsiveness, motor skills, and mood.

Objective 4: To determine if leisure activity participation patterns vary across ages of students and change after two semesters of participation in a fitness program.

Data Collection phase of the study. Timeline Months 1 & 2: Identification of participants, Consents, Baseline data collected (Visit 1) Months 3-9: Fit Club Month 9 (Visit 2) Months 10-12: Summer Break Months13-14: School Start data collection (Visit 3) Months14-18: Data analysis and dissemination

Evaluation/Data Analysis:

Data from students will include factors that affect academic performance, including measures of EF, sensory responsiveness, and motor skills. Physiological statistics such as height and weight will be collected to calculate Body Mass Indices (BMI) for each participant over the course of the study. To achieve the greatest validity, assessments have been selected that obtain the perspectives from several sources: parent/LAR report, teacher report and direct observation. Parent, student, and teacher questionnaires will be administered online. All students, teachers, and parents will be able to use computers with access to the internet. Observation assessments will be conducted by graduate occupational therapy students from the University of Texas Medical Branch. A FitBit® activity tracking wristband with a heart rate monitor and wireless syncing capabilities will be worn by participants and will be used to track resting and peak heart rate, calories burned, steps taken, and sleep quality. Outcome constructs and performance measures are listed below.

Study Outcome: Performance Measure ASD Severity: Social Responsiveness Scale, Second Edition, parent and teacher forms (SRS-2), Sensory Responsiveness: Adolescent/Adult Sensory Profile, Motor Performance: Bruininks-Osteretsky Test of Motor Proficiency, Second Edition (BOT-2), Executive Function: Behavior Rating Inventory of Executive Function, parent and teacher forms (BRIEF), Delis-Kaplan Executive Function System (D-KEFS), Participation: Children's Assessment of Participation and Enjoyment & Preferences for Activities of Children (CAPE/PAC), Life Participation for Parents, Adolescent and Young Adult Activity Card Sort (AYA-ACS), Behavior/Mood: Repetitive Behavior Scale, Depression, Anxiety and Stress Scale (DASS), Effort:Heart Rate and daily steps taken with activity monitoring wristband, Summer Exercise Questionnaire Metabolic Parameters Height and weight scale, Height in inches, Body temperature with no contact thermometer

Significance:

This research has the potential to change policy regarding physical education for students with ASD. If the results of this study show a strong relationship between the level of physical exertion and improvements in factors affecting academic performance, it will suggest adding more physically exerting activities to school curricula for students with ASD. The positive impact of physical exercise has been observed in previous studies, but this study may help to clarify the relationship between effort during exercise and improvements in the factors that support academic performance. The investigators may also gain understanding of the duration and effort of exercise necessary to see improvements in these factors, and whether the benefits are sustained. Examination of regression from non-adherence over the summer will help clarify the necessity of continuous participation. If a relationship is found between effort and the factors supporting academic performance, it will help to better identify options for interventions to improve those factors in students with ASD. Participation data will build a better understanding of leisure activity participation patterns in adolescents with ASD that will help to guide intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 - 18 years
* Diagnosis of ASD
* IQ of 60+, will be provided by Gateway Academy with parental consent
* Willingness to participate in study (i.e. signed assent/consent)
* Conversational use of English language

Exclusion Criteria:

* Dual diagnosis of cerebral palsy or any other major neurologic condition
* Uncorrected hearing or vision problems

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Bruininks-Osteretsky Test of Motor Proficiency, Second Edition | Initial, 9 months
  is a standardized measure of motor proficiency. It generates gender-specific composite subscale scores for: fine manual control, manual coordination, body coordination, strength and agility, and a full motor composite score, and has been normed for children between ages 4 and 21. Participants will be tested at the beginning and end of the school year to detect change in motor proficiency after participating in the intervention.

SECONDARY OUTCOMES:
Change from baseline in Adolescent and Young Adult Activity Card Sort | Initial, 9 months
  is a card sort assessment of participation in everyday activities developed for individuals between the ages of 18-25. It includes activities in categories of obligatory chores, leisure, social, health, wellness or fitness, education and learning, work, and parenting/caring for children. Participants will be tested at the beginning and end of the school year to detect change in activity participation after participating in the intervention.
Change from baseline in Depression, Anxiety and Stress Scale | Initial, 9 months
  is a self-report, 4-point Likert-scale and a quantitative measure of distress along three dimensions: depression, anxiety and stress. Participants will be tested at the beginning and end of the school year to detect change.
Change from baseline in Repetitive Behavior Scale | Initial, 9 months
  An empirically derived parent-reported clinical rating scale for measuring the presence and severity of a variety of forms of restricted, repetitive behaviors that are characteristic of children and adults with Autism Spectrum Disorders (ASD). Six subscales are derived from 43 items consisting of: 1) Stereotyped Behavior, 2) Self-injurious Behavior, 3) Compulsive Behavior, 4) Routine Behavior, 5) Sameness Behavior, and 6) Restricted Behavior. This scale will be administered at the beginning and the end of the school year to detect changes in repetitive behavior from participation in the intervention.
Change from baseline in Sensory Profile Adolescent/Adult | Initial, 9 months
  is a standardized questionnaire for individuals between the ages of 11 and 65, is comprised of 60 statements rated on a Likert (1) never to (5) always scale. Participants will be complete the form at the beginning and end of the school year to detect change in their sensory responsiveness after participating in the intervention.
Change from baseline in Body Mass Indices | Initial, 9 months
  Height and weight will be measured and BMI calculated from that. Height and weight will be measured at the beginning and end of the school year to detect change in BMI after participating in the intervention.
Change from baseline in Exercise Heart Rate | initial, 9 months
  FitbitChargeHR® activity tracking wristband with a HR monitor and wireless syncing capabilities will be worn by participants and will be used to track resting and peak HR. Exercise heart rate will be compared between the beginning and the end of the school year to detect changes after participating in the intervention.
Change from baseline in Delis-Kaplan Executive Function System | Initial, 9 months
  is the first nationally standardized set of tests to evaluate higher level cognitive. Participants will be tested at the beginning and end of the school year to detect change in executive function after participating in the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia L Hilton, PhD, Principal Investigator — University of Texas
Locations (1):
- Gateway Academy, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No